CLINICAL TRIAL: NCT01664182
Title: A Randomized Phase 2 Study of AMG 386 With or Without Continued Anti-Vascular Endothelial Growth Factor (VEGF) Therapy in Patients With Renal Cell Carcinoma Who Have Progressed on Bevacizumab, Pazopanib, Sorafenib, or Sunitinib
Brief Title: Trebananib With or Without Bevacizumab, Pazopanib Hydrochloride, Sorafenib Tosylate, or Sunitinib Malate in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01289; NCI-2012-01289 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-122; P9048_A12PAMDREVW01; CDR0000738785; 9048 (Other: City of Hope Comprehensive Cancer Center); 9048 (Other: CTEP); N01CM00038 (NIH); P30CA033572 (NIH)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Advanced Renal Cell Carcinoma; Advanced Sarcomatoid Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Immunoglobulin G; Disulfides; pazopanib; Sorafenib; Sunitinib; trebananib

ARMS (2):
- Arm I (trebananib monotherapy) (Experimental): Patients receive trebananib IV over 30-60 minutes on days 1, 8, 15, 22, 29, and 36. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Trebananib
- Arm II (trebananib and anti-VEGF therapy) (Experimental): Patients receive trebananib as in Arm I and either bevacizumab IV over 30-90 minutes on days 1, 15, and 29, pazopanib hydrochloride PO QD on days 1-42, sorafenib tosylate PO BID on days 1-42, or sunitinib malate PO QD on days 1-28. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Pazopanib Hydrochloride; Drug: Sorafenib Tosylate; Drug: Sunitinib Malate; Biological: Trebananib

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
  Arms: Arm II (trebananib and anti-VEGF therapy)
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
  Arms: Arm II (trebananib and anti-VEGF therapy)
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
  Arms: Arm II (trebananib and anti-VEGF therapy)
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent
  Arms: Arm II (trebananib and anti-VEGF therapy)
Biological: Trebananib — Given IV
  Other Names: AMG 386; AMG386; Angiopoietin 1/2-Neutralizing Peptibody AMG 386

SUMMARY:
This randomized phase II trial studies how well trebananib with or without bevacizumab, pazopanib hydrochloride, sorafenib tosylate, or sunitinib malate works in treating patients with kidney cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Trebananib may stop the growth of tumor cells by blocking blood flow to the tumor. Immunotherapy with monoclonal, such as bevacizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Pazopanib hydrochloride, sorafenib tosylate, and sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. It is not yet known whether giving trebananib with or without bevacizumab, pazopanib hydrochloride, sorafenib tosylate, or sunitinib malate is more effective in treating kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the overall response rate (complete response [CR] + partial response [PR]) of trebananib (AMG 386) alone and in combination with continuation of previously administered bevacizumab, pazopanib hydrochloride (pazopanib), sorafenib tosylate (sorafenib), or sunitinib malate (sunitinib) in advanced renal cell carcinoma.

SECONDARY OBJECTIVES:

I. To evaluate progression free survival in each arm. II. To evaluate the tolerance and toxicity of AMG 386 alone and in combination with continuation of the prior VEGF targeted agent.

CORRELATIVE OBJECTIVES:

I. To evaluate the association between pretreatment tumor gene expression levels and response to AMG 386 in combination with continuation of the prior VEGF targeted agent.

II. To evaluate the association between single nucleotide polymorphisms (SNPs) in angiogenic genes and response to AMG 386 in combination with continuation of the prior VEGF targeted agent.

III. To compare changes in circulating angiogenic factors in patients treated with AMG 386 monotherapy to those treated with AMG 386 in combination with VEGF-targeted therapy.

IV. To compare expression of angiogenic genes from archival tumor specimens to the expression in biopsy specimens obtained after progression on anti-VEGF therapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive trebananib intravenously (IV) over 30-60 minutes on days 1, 8, 15, 22, 29, and 36. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive trebananib as in Arm I and either bevacizumab IV over 30-90 minutes on days 1, 15, and 29, pazopanib hydrochloride orally (PO) once daily (QD) on days 1-42, sorafenib tosylate PO twice daily (BID) on days 1-42, or sunitinib malate PO QD on days 1-28. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed renal cell carcinoma except medullary or collecting duct subtypes; sarcomatoid differentiation will be allowed
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have documented radiologic or clinical progressive disease following at least one prior anti-VEGF regimen administered either as a single agent or in combination with other agents for at least 8 weeks; the prior anti-VEGF treatment regimen must have included bevacizumab, pazopanib, sorafenib or sunitinib administered not more than 12 weeks before study entry; Note: enrollment not more than 8 weeks after the last dose of anti-VEGF therapy is encouraged; nevertheless, intercurrent therapy with an mTOR inhibitor (everolimus or temsirolimus) will be allowed if progression on that treatment is observed within 12 weeks of the prior anti-VEGF therapy
* Any number of prior regimens is allowed; prior investigational therapy is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< institutional upper limits of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) =< upper limit of normal (ULN) per institutional laboratory range
* International normalized ratio (INR) =< 1.5
* Creatinine within normal institutional limits OR creatinine clearance > 40 mL/min per 24 hour (h) urine collection or calculated according to the Cockcroft-Gault formula
* Urinary protein =< 100 mg/dL in urinalysis or =< 1+ on dipstick, unless quantitative protein is < 1000 mg in a 24 h urine sample
* Generally well-controlled blood pressure with systolic blood pressure =< 140 mmHg AND diastolic blood pressure =< 90 mmHg prior to enrollment; the use of anti-hypertensive medications to control hypertension is permitted
* Patients must have a tumor site amenable to biopsy as determined by the treating investigator; any questions regarding suitability of a site for biopsy will be adjudicated by the principal investigator
* Patients must be willing to consent to tumor biopsy for research purposes
* Patients should have archival tumor tissue (either unstained slides or tumor blocks) available for retrieval
* The effects of AMG 386 are known to be detrimental to fetal development; for this reason and because inhibitors of angiogenesis as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 6 months after completion of AMG 386; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of AMG 386 and bevacizumab, pazopanib, sunitinib, or sorafenib administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Intolerance of prior treatment with bevacizumab, pazopanib, sorafenib, or sunitinib; Note: subjects who required a dose reduction of pazopanib, sorafenib, or sunitinib during prior therapy MAY be eligible if they tolerated the agent after dose level reduction (to a minimum of dose level -2 as defined in this protocol)
* Central nervous system metastases unless: (1) metastases have been treated and have remained controlled for at least two weeks following treatment, AND (2) patient has no residual neurological dysfunction off corticosteroids for at least one week; a CT or MRI to evaluate for central nervous system (CNS) disease is required for symptomatic patients only
* History of venous or arterial thromboembolism within 12 months prior to enrollment/randomization
* History of clinically significant bleeding within 6 months of enrollment/randomization
* Unresolved toxicities from prior systemic therapy that are Common Terminology Criteria in Adverse Events (CTCAE) version 3.0 or 4.0 >= grade 2 in severity except alopecia
* Currently or previously treated with AMG 386, or other molecules that inhibit the angiopoietins or Tie2 receptor
* Clinically significant cardiovascular disease within 12 months prior to enrollment/randomization, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication or placement of percutaneous transluminal coronary angioplasty/stent
* Major surgery within 28 days prior to enrollment or still recovering from prior surgery
* Minor surgical procedures except placement of tunneled central venous access device within 3 days prior to enrollment
* Non-healing wound, ulcer (including gastrointestinal), or fracture
* Subject not consenting to the use of highly effective contraceptive precautions (e.g., double barrier method [i.e., condom plus diaphragm]) during the course of the study and for 6 months after administration of the last study medication
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AMG 386 or the anti-VEGF agent used in study
* History of allergic reactions to bacterially-produced proteins
* Patients who have had anti-VEGFR tyrosine kinase inhibitor within 1 week, mTOR inhibitor within 1 week or anti-VEGF antibody therapy within 3 weeks prior to entering the study; patients who have had other forms of chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have not yet completed at least 21 days (30 days for prior monoclonal antibody therapy) since ending other investigational device or drug trials, or who are currently receiving other investigational treatments
* Patients receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP450 3A4) are ineligible; caution is advised for patients requiring weak or moderate CYP450 3A4 inhibitors or inducers; specifically prohibited medicines include indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, carbamazepine, phenobarbital, phenytoin, pioglitazone, rifabutin, rifampin, St. John's wort, and troglitazone
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because AMG 386, bevacizumab, pazopanib, sorafenib, and sunitinib are inhibitors of angiogenesis with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AMG 386, breastfeeding must be discontinued if the mother is treated with AMG 386
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pazopanib, sorafenib, or sunitinib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Inability to take oral medications on a continuous basis; patients who are to take pazopanib, sorafenib, or sunitinib and are unable to swallow pills whole are ineligible (the pills cannot be crushed or broken)
* Any condition which in the investigator's opinion makes the subject unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Semrad, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (12):
- United States (12):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - VCU Massey Cancer Center at Hanover Medical Park, Mechanicsville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Trebananib Monotherapy) | Arm II (Trebananib and Anti-VEGF Therapy)
Started | 19 | 22
Completed | 17 | 18
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Trebananib Monotherapy) | Arm II (Trebananib and Anti-VEGF Therapy) | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Median (Full Range); unit: years] | 64 [49 to 76] | 59 [46 to 74] | 60 [46 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 2 | 0 | 2
  Asian/Pacific Islander | 0 | 1 | 1
  Black | 2 | 1 | 3
  Hispanic | 4 | 4 | 8
  White | 9 | 12 | 21
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35
ECOG Performance Score [Count of Participants; unit: Participants] — ECOG (Eastern Cooperative Oncology Group) Performance Score is a measure of patients' ability to tolerate therapies in serious illness, e.g. chemotherapy.
  0 = Asymptomatic: Fully active, able to carry on all pre-disease activities without restriction
  1. = Restricted in strenuous activity, ambulatory and able to do light work
  2. = Capable of all self care, but no work activities; out of bed > 50% of day
  3. = Capable of limited self-care; confined to bed or chair > 50% of day
  4. = Completely disabled; no self-care; confined to bed or chair
  5. = Dead
  Participants
    0 | 12 | 11 | 23
    1 | 5 | 7 | 12
Prior Anti-VEGF Agent [Count of Participants; unit: Participants] — anti-VEGF agent: anti-Vascular Endothelial Growth Factor receptor agent.
  Participants
    Bevacizumab | 5 | 10 | 15
    Pazopanib | 6 | 5 | 11
    Sorafenib | 2 | 2 | 4
    Sunitinib | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Observed Response Rate
Description: Defined as the total number of efficacy-evaluable patients who achieve a complete or partial response by RECIST version 1.1 criteria, assessed by MRI: Complete Response (CR), Disappearance of all target lesions:
  any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Best response will be listed for each patient and summarized using standard descriptive methods-point estimate and associated confidence intervals.
Time Frame: Up to 8 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients responding
Arm/Group | Arm I (Trebananib Monotherapy) | Arm II (Trebananib and Anti-VEGF Therapy)
Number analyzed (Participants) | 17 | 18
percentage of patients responding | 0 [0 to 20] | 11 [1 to 35]

2. Primary Outcome: Tumor Response
Description: Tumor Response Classification
Time Frame: at 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Trebananib Monotherapy) | Arm II (Trebananib and Anti-VEGF Therapy)
Number analyzed (Participants) | 17 | 18
Participants
  Partial Response | 0 | 2
  Stable Disease | 5 | 8
  Progressive Disease | 11 | 6
  Not Evaluable | 1 | 2

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Time to reach Kaplan-Meier median survival (outcome being death or progression) (95% Confidence Interval) is reported. Progressive Disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered a progression.)
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 8 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Trebananib Monotherapy) | Arm II (Trebananib and Anti-VEGF Therapy)
Number analyzed (Participants) | 17 | 18
months | 2.7 [2.3 to 4.7] | 5.2 [2.7 to 10.8]

4. Secondary Outcome: Number of Participants With Grade 3, 4, 5 Toxicities Related to the Treatment Drugs
Description: Adverse events were graded using CTCAE version 5.0. Grades 3, 4, 5 (on a scale of 1 to 5, 5 being the worst grade - death) toxicities related ('Possibly', 'Probably', or 'Definitely') to the treatment drugs (AMG 386 alone or in combination with prior VEGF targeted agent).
Time Frame: 8 weeks for adverse events. Until removal from the study or to death for late adverse events, up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Trebananib Monotherapy) | Arm II (Trebananib and Anti-VEGF Therapy)
Number analyzed (Participants) | 17 | 18
Participants
  SAE Cardiac disorders: Cardiac arrest | 0 | 1
  SAE Metabolism and nutrition disorders: Hypokalemia | 1 | 0
  SAE Respiratory, thoracic and mediastinal disorders: Dyspnea | 1 | 1
  SAE Respiratory, thoracic and mediastinal disorders: Pleural effusion | 1 | 0
  Blood and lymphatic system disorders: Anemia | 0 | 1
  General disorders and administrative site conditions: Fatigue | 1 | 3
  Investigations: Lymphocyte count decreased | 0 | 1
  Investigations: Weight gain | 0 | 1
  Metabolism and nutrition disorders: Acidosis | 0 | 1
  Metabolism and nutrition disorders: Hyperglycemia | 1 | 0
  Metabolism and nutrition disorders: Hyponatremia | 0 | 1
  Musculoskeletal and connective tissue disorders: Back pain | 1 | 1
  Vascular disorders: Hypertension | 3 | 3

5. Other Pre Specified Outcome: Changes in Circulating Angiogenic Factors
Description: Analyzed as continuous variables (most likely after transformation). The gene expression results from the pretreatment tumor biopsies are expressed as ratios between that of the gene of interest and the internal reference gene beta-actin and can be analyzed as continuous variables - generally after log transformation.
Time Frame: Baseline to up to 8 weeks
Population: availability of samples. attrition from the study.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm I (Trebananib Monotherapy) | Arm II (Trebananib and Anti-VEGF Therapy)
Number analyzed (Participants) | 17 | 18
pg/ml
  Angiopoietin--2 at baseline: number analyzed (Participants) | 15 | 15
  Angiopoietin--2 at baseline | 3909 [3246 to 4863] | 3237 [2424 to 4813]
  Angiopoietin--2 prior to cycle 2: number analyzed (Participants) | 14 | 15
  Angiopoietin--2 prior to cycle 2 | 132156 [110775 to 160316] | 120956 [84474 to 131643]
  Angiopoietin--2 prior to cycle 3: number analyzed (Participants) | 9 | 11
  Angiopoietin--2 prior to cycle 3 | 125928 [114871 to 141528] | 96075 [84200 to 150486]
  Tie--2 at baseline: number analyzed (Participants) | 15 | 15
  Tie--2 at baseline | 803 [510 to 1035] | 835 [650 to 1094]
  Tie--2 prior to cycle 2: number analyzed (Participants) | 14 | 15
  Tie--2 prior to cycle 2 | 783 [535 to 1041] | 671 [571 to 856]
  Tie--2 prior to cycle 3: number analyzed (Participants) | 9 | 11
  Tie--2 prior to cycle 3 | 912 [263 to 1232] | 753 [424 to 912]
  VEGF--A at baseline: number analyzed (Participants) | 15 | 15
  VEGF--A at baseline | 27.3 [10.5 to 48.4] | 26.1 [19.6 to 38.0]
  VEGF--A prior to cycle 2: number analyzed (Participants) | 14 | 15
  VEGF--A prior to cycle 2 | 21.3 [10.5 to 29.0] | 33.4 [13.6 to 48.2]
  VEGF--A prior to cycle 3: number analyzed (Participants) | 9 | 11
  VEGF--A prior to cycle 3 | 20.7 [0.3 to 34.2] | 41.2 [26.1 to 56.7]
  PIGF at baseline: number analyzed (Participants) | 15 | 15
  PIGF at baseline | 31.1 [26.1 to 35.2] | 30.7 [28.3 to 46.7]
  PIGF prior to cycle 2: number analyzed (Participants) | 14 | 15
  PIGF prior to cycle 2 | 30.5 [21.8 to 36.0] | 33.6 [29.9 to 39.2]
  PIGF prior to cycle 3: number analyzed (Participants) | 9 | 11
  PIGF prior to cycle 3 | 31.4 [30.5 to 34.3] | 31.5 [26.3 to 41.8]
  VEGFR--3 at baseline: number analyzed (Participants) | 15 | 15
  VEGFR--3 at baseline | 873 [157 to 1073] | 489 [50 to 898]
  VEGFR--3 prior to cycle 2: number analyzed (Participants) | 14 | 15
  VEGFR--3 prior to cycle 2 | 722 [117 to 869] | 50 [50 to 321]
  VEGFR--3 prior to cycle 3: number analyzed (Participants) | 9 | 11
  VEGFR--3 prior to cycle 3 | 489 [362 to 954] | 50 [50 to 416]
  VEGF--C at baseline: number analyzed (Participants) | 15 | 15
  VEGF--C at baseline | 255 [72 to 425] | 283 [251 to 380]
  VEGF--C prior to cycle 2: number analyzed (Participants) | 14 | 15
  VEGF--C prior to cycle 2 | 209 [67 to 340] | 311 [247 to 357]
  VEGF--C prior to cycle 3: number analyzed (Participants) | 9 | 11
  VEGF--C prior to cycle 3 | 230 [45 to 358] | 311 [154 to 503]
  IL--8 at baseline: number analyzed (Participants) | 15 | 15
  IL--8 at baseline | 0.1 [0.1 to 12.6] | 0.1 [0.1 to 4.0]
  IL--8 prior to cycle 2: number analyzed (Participants) | 14 | 15
  IL--8 prior to cycle 2 | 3.6 [0.1 to 17.5] | 5.9 [0.1 to 13.5]
  IL--8 prior to cycle 3: number analyzed (Participants) | 9 | 11
  IL--8 prior to cycle 3 | 2.5 [0.1 to 8.1] | 0.4 [0.1 to 17.3]
  ICAM--1 at baseline: number analyzed (Participants) | 15 | 15
  ICAM--1 at baseline | 161879 [103645 to 240620] | 243594 [185653 to 601003]
  ICAM--1 prior to cycle 2: number analyzed (Participants) | 14 | 15
  ICAM--1 prior to cycle 2 | 193335 [117584 to 247434] | 239027 [160295 to 318968]
  ICAM--1 prior to cycle 3: number analyzed (Participants) | 9 | 11
  ICAM--1 prior to cycle 3 | 262636 [221161 to 266594] | 200959 [150610 to 276615]
  VCAM--1 at baseline: number analyzed (Participants) | 15 | 15
  VCAM--1 at baseline | 965554 [738499 to 1421550] | 1307900 [982643 to 1946700]
  VCAM--1 prior to cycle 2: number analyzed (Participants) | 14 | 15
  VCAM--1 prior to cycle 2 | 1336300 [955663 to 1903550] | 1850000 [1327000 to 2555600]
  VCAM--1 prior to cycle 3: number analyzed (Participants) | 9 | 11
  VCAM--1 prior to cycle 3 | 982488 [969237 to 1581000] | 1666200 [1351500 to 2091050]
  FGF2 at baseline: number analyzed (Participants) | 15 | 15
  FGF2 at baseline | 124 [105 to 136] | 120 [105 to 136]
  FGF2 prior to cycle 2: number analyzed (Participants) | 14 | 15
  FGF2 prior to cycle 2 | 112 [89 to 131] | 110 [95 to 132]
  FGF2 prior to cycle 3: number analyzed (Participants) | 9 | 11
  FGF2 prior to cycle 3 | 131 [104 to 136] | 120 [97 to 133]
  PDGF -- AA at baseline: number analyzed (Participants) | 15 | 15
  PDGF -- AA at baseline | 351 [237 to 788] | 478 [112 to 647]
  PDGF -- AA prior to cycle 2: number analyzed (Participants) | 14 | 15
  PDGF -- AA prior to cycle 2 | 291 [190 to 394] | 262 [213 to 829]
  PDGF -- AA prior to cycle 3: number analyzed (Participants) | 9 | 11
  PDGF -- AA prior to cycle 3 | 264 [119 to 710] | 173 [105 to 777]
Statistical Analysis 1: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); Arm A vs Arm B shift test on Angiopoietin -- 2 prior to cycle 2. Wilcoxon rank-sum test p-value; Test type: Other — Two sided hypothesis. Wilcoxon rank-sum test comparing the two arms in terms of the ratio of the post-treatment levels divided by the baseline; p = 0.86, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. A-priori threshold for statistical significance is 0.05
Statistical Analysis 2: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); Angiopoietin -- 2 prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.76, Wilcoxon (Mann-Whitney) — Angiopoietin -- 2 prior to cycle 3
Statistical Analysis 3: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); Tie--2 Prior to cycle 2; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.14, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparison. A-priori threshold for statistical significance is 0.05
Statistical Analysis 4: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); Tie -- 2 prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.069, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. A-priori threshold for statistical significance is 0.05
Statistical Analysis 5: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); VEGF -- A prior to cycle 2; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.19, Wilcoxon (Mann-Whitney) — P-value is not adjusted for multiple comparisons. A-priori threshold for statistical significance is 0.05
Statistical Analysis 6: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); VEGF--A prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.046, Wilcoxon (Mann-Whitney) — P-value is not adjusted for multiple comparisons. The a-priori threshold for statistical significance is 0.05
Statistical Analysis 7: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); PIGF Prior to Cycle 2; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.029, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons. A-priori threshold for statistical significance is 0.05
Statistical Analysis 8: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); PIGF prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.20, Wilcoxon (Mann-Whitney) — P-value is not adjusted for multiple comparisons. A priori threshold for statistical significance is 0.05
Statistical Analysis 9: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); VEGFR--3 prior to cycle 2; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.11, Wilcoxon (Mann-Whitney) — The p-value was not adjusted for multiple comparisons. The a-priori threshold for statistical significance is 0.05
Statistical Analysis 10: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); VEGFR--3 prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.068, Wilcoxon (Mann-Whitney) — P-value was not adjusted for multiple comparisons. The a-priori threshold for statistical significance was 0.05
Statistical Analysis 11: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); VEGF--C prior to cycle 2; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.61, Wilcoxon (Mann-Whitney) — The p-value was not adjusted for multiple comparisons. The a-priori threshold for statistical significance was 0.05
Statistical Analysis 12: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); VEGF--C prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.27, Wilcoxon (Mann-Whitney) — Two sided hypothesis. Wilcoxon rank-sum test comparing the two arms in terms of the ratio of the post-treatment levels divided by the baseline
Statistical Analysis 13: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); IL--8 prior to cycle 2; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.61, Wilcoxon (Mann-Whitney) — The p-value was not adjusted for multiple comparisons. The a-priori threshold for statistical significance was 0.05
Statistical Analysis 14: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); IL--8 prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.49, Wilcoxon (Mann-Whitney) — The p-value was not adjusted for multiple comparisons, and the a-priori threshold for statistical significance was 0.05
Statistical Analysis 15: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); ICAM--1 prior to cycle 2; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.82, Wilcoxon (Mann-Whitney) — The p-value was not adjusted for multiple comparisons. The a-priori threshold for statistical significance was 0.05
Statistical Analysis 16: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); ICAM--1 prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.069, Wilcoxon (Mann-Whitney) — The p-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05
Statistical Analysis 17: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); VCAM--1 prior to cycle 2; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.34, Wilcoxon (Mann-Whitney) — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05
Statistical Analysis 18: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); VCAM--1 prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.046, Wilcoxon (Mann-Whitney) — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was set to 0.05
Statistical Analysis 19: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); FGF2 prior to cycle 2; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.11, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 18]
Statistical Analysis 20: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); FGF2 prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.23, Wilcoxon (Mann-Whitney) — The p-value was adjusted for multiple comparisons. The a prior threshold for statistical significance was set to 0.05
Statistical Analysis 21: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); PDGF--AA prior to cycle 2; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.37, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 18]
Statistical Analysis 22: Comparison: Arm I (Trebananib Monotherapy) vs Arm II (Trebananib and Anti-VEGF Therapy); PDGF--AA prior to cycle 3; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.35, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 18]

ADVERSE EVENTS:
Time Frame: 8 weeks for adverse events. Until removal from the study or to death for late adverse events, up to 12 weeks
Description: CTCAE version 4.0 will be used until March 31, 2018. CTCAE version 5.0 will be used from April 1, 2018.
Arm/Group | Arm I (Trebananib Monotherapy) | Arm II (Trebananib and Anti-VEGF Therapy)
All-Cause Mortality (participants affected / at risk) | 0/17 | 2/18
Serious Adverse Events (participants affected / at risk) | 10/17 | 18/18
Other Adverse Events (participants affected / at risk) | 16/17 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Trebananib Monotherapy) (N=17) | Arm II (Trebananib and Anti-VEGF Therapy) (N=18)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Suspected pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Trebananib Monotherapy) (N=17) | Arm II (Trebananib and Anti-VEGF Therapy) (N=18)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Decreased RBC count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 3 (3)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Blurred vision (Eye disorders) | 4 (4) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 2 (2)
redness (Eye disorders) | 0 (0) | 1 (1)
Solitary Diverticulm in Caecum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Dry heaves (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 8 (8)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
belching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrophic Dermatitis (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 2 (2)
Claudication (General disorders) | 1 (1) | 0 (0)
Decreased Monocytes (General disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 3 (3) | 5 (5)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (9) | 10 (10)
Fever (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Hypoproteinemia (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0)
Leucocytes in urine (General disorders) | 1 (1) | 0 (0)
Leukocytes in urine (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 2 (2) | 2 (2)
Rash (General disorders) | 0 (0) | 1 (1)
general edema (General disorders) | 0 (0) | 1 (1)
generalised edema (General disorders) | 0 (0) | 1 (1)
high triglycerides (General disorders) | 1 (1) | 0 (0)
increased Urobilinogen (General disorders) | 0 (0) | 1 (1)
sweaty (General disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Epididymidis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Cellulitis of left hand (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Cholesterol high (Investigations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 4 (4) | 10 (10)
Hemoglobin increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 4 (4)
Weight gain (Investigations) | 2 (2) | 6 (6)
Weight loss (Investigations) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 4 (4)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 6 (6) | 7 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Gout flare (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
left rotator cuff tendinitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
neurogenic claudication (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
right shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 5 (5)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
jerking sensation (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 4 (4) | 7 (7)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
urinary hesitancy (Renal and urinary disorders) | 0 (0) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Epidermoid cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 11 (11)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT01664182/Prot_SAP_000.pdf